CLINICAL TRIAL: NCT02655991
Title: Homecoming Line: Telephone Support for Veterans
Acronym: HCL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Collaborators: Durham VA Medical Center (U.S. Federal Agency); VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Craig S. Rosen, Ph.D., Deputy Director, National Center for PTSD, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: W81XWH=08-2-0096
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Stress Disorders, Post-Traumatic; Ambulatory Care; Telemedicine; Remote Consultation; Health Services Accessibility
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telephone Case Monitoring (Experimental): Telephone care management augmenting treatment as usual
  Interventions: Behavioral: Telephone Case Monitoring; Behavioral: Treatment as Usual
- Treatment as Usual (Active Comparator): Case management, psychotherapy, and pharmacotherapy as usual
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Telephone Case Monitoring — Outpatient mental health treatment as usual (normal case management, psychotherapy and/or pharmacotherapy) augmented by up to six fortnightly telephone monitoring and support calls from a case manager during the first three months of treatment.
  Arms: Telephone Case Monitoring
Behavioral: Treatment as Usual — Outpatient mental health treatment as usual (normal case management, psychotherapy and/or pharmacotherapy).

SUMMARY:
This study will determine whether telephone support improves clinical outcomes of veterans who begin outpatient treatment for posttraumatic stress disorder. Participants will be randomly assigned to receive either usual care or usual care supplemented by biweekly monitoring and support by telephone during the first 3 months of treatment. Patients in both conditions will be compared on PTSD symptoms, engagement in treatment, violence and drinking at 4 months and 12 months after entering treatment.

DETAILED DESCRIPTION:
This multisite randomized controlled trial will test whether a 3-month period of providing telephone monitoring to PTSD patients as a supplement to usual specialty mental health care improves 12-month clinical outcomes (a reduction in PTSD symptoms, violence, and substance use). Secondarily, this study will determine whether telephone monitoring promotes better engagement in outpatient treatment (Number of mental health and psychotherapy visits during the 3-month intervention period).

Demand for VA PTSD treatment is increasing as troops return from combat deployments in Afghanistan and Iraq. Telemedicine is likely to be an important component in developing more effective and efficient models of PTSD care that improves patient functioning and treatment utilization. It is hoped that using telephone case monitoring as an inexpensive adjunct to standard care may improve clinical outcomes and reduce hospitalization among veterans with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* VA patients newly entering outpatient treatment mental health treatment for PTSD starting a new phase of outpatient PTSD treatment (e.g., transitioning from a psycho-education group to active psychotherapy) at one of the study sites.

Exclusion Criteria:

* Active duty personnel
* Cognitive impairment which precludes giving informed consent
* Initiating residential or inpatient treatment rather than outpatient treatment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2008-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist (PCL) Slope | 12 months
  Slope of improvement on the PTSD Checklist, a self-report measure of PTSD symptoms.

SECONDARY OUTCOMES:
PTSD psychotherapy visits - intervention period | 3 months
  Number of psychotherapy visits for PTSD (psychotherapy procedure code + PTSD diagnosis code) completed during the 3 month intervention period.
Other mental health visits - intervention period | 3 months
  Number of "other" mental health visits (mental health visits without psychotherapy procedure code and/or without a PTSD diagnosis code) completed during the 3 month intervention period.
Depression slope | 12 months
  Slope of improvement on the Center for Epidemiological Studies Scale, a self-report measure of depression symptoms.
Alcohol problems slope | 12 months
  Slope of improvement on the Addiction Severity Index Alcohol Composite, a self-report measure of alcohol-related problems.
Drug problems slope | 12 months
  Slope of improvement on the Addiction Severity Index Drug Composite, a self-report measure of drug-related problems.
Aggression slope | 12 months
  Slope of improvement on a six-item self-report measure of aggressive behaviors, adapted from the Conflict Tactics Scale.
Quality of Life slope | 12 months
  Slope of improvement on a self-report quality measure used in the Veterans Affairs Military Stress Treatment Assessment study.
PTSD psychotherapy visits -- follow-up period | months 4-12
  Number of psychotherapy visits for PTSD (psychotherapy procedure code + PTSD diagnosis code) completed during the post-intervention period (months 4-12).
Other mental health visits -- follow-up period | months 4-12
  Number of "other" mental health visits (mental health visits without psychotherapy procedure code and/or without a PTSD diagnosis code) completed during the post-intervention period (months 4-12).
Selective serotonin reuptake inhibitor refills (medication possession ratio) | 12 months
  Number of days' supply of selective serotonin reuptake inhibitors (SSRIs) obtained divided by 365 days.
Prazosin refills (medication possession ratio) | 12 months
  Number of days' supply of Prazosin obtained divided by 365 days.

CONTACTS AND LOCATIONS:
Overall Officials: Craig S. Rosen, Ph.D., Principal Investigator — VA Palo Alto Health Care System
Locations (3):
- United States (3):
  - VA Palo Alto Health Care System (Meno Park Division), Menlo Park, California
  - Durham VA Medical Center, Durham, North Carolina
  - VA Puget Sound Health Care System (American Lake), Lakewood, Washington

REFERENCES:
- [Derived] Rosen CS, Azevedo KJ, Tiet QQ, Greene CJ, Wood AE, Calhoun P, Bowe T, Capehart BP, Crawford EF, Greenbaum MA, Harris AH, Hertzberg M, Lindley SE, Smith BN, Schnurr PP. An RCT of Effects of Telephone Care Management on Treatment Adherence and Clinical Outcomes Among Veterans With PTSD. Psychiatr Serv. 2017 Feb 1;68(2):151-158. doi: 10.1176/appi.ps.201600069. Epub 2016 Oct 17. PMID 27745535